CLINICAL TRIAL: NCT04106206
Title: Multiple-Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study of LY3372689
Brief Title: A Safety Study of LY3372689 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17242; I9X-MC-MTAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3372689 (Experimental): LY3372689 administered orally
  Interventions: Drug: LY3372689
- Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3372689 — Administered orally
  Arms: LY3372689
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This study is being conducted to determine the safety profile of the study drug after it is given by mouth to healthy participants. Blood tests will be performed to check how much LY3372689 gets into the bloodstream and how long the body takes to get rid of it. Each enrolled participant will receive multiple doses of LY3372689 or placebo and will remain in the study for up to eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy vasectomized male or a female who cannot get pregnant
* Have a body mass index (BMI) of 18.5 to ≤30 kilograms per square meter (kg/m²)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG, heart tracing), blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for ease of blood sampling

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Smoke more than the equivalent of 10 cigarettes per day and are unwilling to stop smoking for study procedure
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate or could interfere with understanding the results of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Observed by the Investigator During Study Drug Administration | Baseline through final follow-up at approximately Day 30
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3372689 | Day 1 postdose through Day 15
  PK: Cmax of LY3372689
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3372689 | Day 1 postdose through Day 15
  PK: AUC of LY3372689

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No